CLINICAL TRIAL: NCT06692218
Title: Leadless Pacemaker Implantation Positions and Its Relationship with Procedure Efficacy and Complication
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tam Tsz Kin, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Leadless-CT study
Record Dates: First submitted 2024-09-26; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Leadless Pacemaker
Keywords: Leadless pacemaker

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CT (Other): All patients will have a non-contrast, ECG-gated CT heart to adjudicate implant position of leadless pacemaker.
  Interventions: Device: Leadless pacemaker

INTERVENTIONS:
Device: Leadless pacemaker — Patients who will implant leadless pacemakers or already implanted leadless pacemakers since 1 Jan 2015 will be recruited. After the implantation, patients will be invited back for a noncontrast, ECG-gated CT heart. It will be timed at the end diastole and a 3D reconstruction will be performed.

SUMMARY:
Leadless pacemakers (LP) are safe and effective alternatives to transvenous pacemakers in select patients. Advances in battery and electronics technology allow for the entire pacemaker system to be implanted into the right ventricle, bypassing many of the weaknesses of transvenous pacemakers. Traditionally leadless pacemakers have been implanted in the right ventricular (RV) septum to prevent cardiac perforation, and much emphasis is placed during implantation to ensure a septal implant. However, in Asians with smaller heart sizes, septal implantation may be unfeasible. Cases of RV free wall implant have been achieved without any complications. This study aims to examine patients previously implanted with LP and determine their final attachment location. If a substantial portion of complication-free patients had RV free wall implants, then it can be argued the additional effort to ensure a septal implant is unnecessary. Additionally, intraoperative data, such as the intracardiac electrogram, may contain parameters correlated with implant position. This study also aims to study this correlation to guide future implant procedures.

This is a prospective-retrospective cohort study. Patients who will implant leadless pacemakers or already implanted leadless pacemakers since 1 Jan 2015 will be recruited. After the implantation, patients will be invited back for a noncontrast ECG-gated CT heart. It will be timed at the end diastole and a 3D reconstruction will be performed. The attachment of the leadless pacemaker to the RV will be adjudicated from the CT. The patients' pre-operative laboratory tests, baseline demographics, medical history, LP electrical data and pre- and post-operative medication regiment will be collected retrospectively from their medical records in the Hospital Authority's Clinical Management System (CMS) and Clinical Data Analysis and Reporting System (CDARS).

ELIGIBILITY:
Inclusion Criteria:

* Patients who will implant leadless pacemaker or already implanted leadless pacemaker since 1 Jan 2015
* Patients with ability to provide informed consent

Exclusion Criteria:

* Patients who cannot provide informed consent
* Patient < 18 years old
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Location of leadless pacemaker implantation | From date of enrollment to date of CT or echocardiogram, up to 1 year
  Determine the exact location of leadless pacemaker implantation

SECONDARY OUTCOMES:
Implant location prediction with electrical parameters | From date of enrollment to date of CT or echocardiogram, up to 1 year
  Correlate leadless pacemaker electrical parameters (including electrogram characteristics, pacing threshold and sensing) to leadless pacemaker implant position (septal, apex or free wall).

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong